CLINICAL TRIAL: NCT02443415
Title: Acute and Long-term Neuroanatomical and Cognitive Evaluation of Adult Patients With First and Recurrent Episodes of Diabetic Ketoacidosis
Brief Title: Diabetic Ketoacidosis: Brain Morphology and Cognition
Acronym: DKA-Cog
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Other Study IDs: IRB00077046
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Healthy Controls: Non-diabetic subjects
- Diabetics without DKA: Diabetic subjects (recent(< 1 year) diagnosis of diabetes) without a history of diabetic ketoacidosis (DKA)
- First episode of DKA: Diabetic subjects that just had their primary event of diabetic ketoacidosis (DKA)
- Three or more DKA episodes: Diabetic subjects who have had three or more diabetic ketoacidosis (DKA) episodes

SUMMARY:
The purpose of this study is to assess brain and memory changes in patients with uncontrolled diabetes (a condition called diabetic ketoacidosis (DKA))

DETAILED DESCRIPTION:
Diabetic ketoacidosis (DKA) is a common and serious medical problem. Most cases occur when patients forget or stop insulin injections. Some patients require frequent admissions to the hospital with DKA after stopping insulin. Many patients do not know why they stop insulin therapy. The investigators will test if patients with one or more episodes of DKA have poor memory and brain changes that may lead to poor management.

In this study, the investigators will perform memory testing and brain images in subjects with initial DKA episode and subjects with more than 3 episodes of DKA. The results will be compared to subjects with diabetes and no history of DKA and healthy (non-diabetic) subjects. Each subject with DKA will have an MRI and cognitive testing done shortly after hospital discharge, 1 month, and 3 months after hospital discharge. Diabetic subjects without DKA and healthy controls will only come in for a single baseline visit and have a MRI and cognitive testing done.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes with diabetic ketoacidosis (DKA)
* Age 18-50 years
* Newly diagnosed or history of noncompliance with insulin therapy as precipitating cause of DKA
* No significant medical or surgical illness as precipitating cause of DKA

Exclusion Criteria:

* Significant medical/surgical illness as precipitating cause of DKA (i.e. myocardial infarction, major surgery)
* Associated significant medical or surgical condition within 6 months history
* History of hypoglycemia unawareness
* History of seizures, ischemic stroke or hemorrhage, and severe head trauma
* History of symptomatic stenosis of major intracranial vessels
* Dementia (mini-mental state examination (MMSE) score (r ≤ 24) or inability to cooperate)
* Liver or renal failure or transplant
* Severe hypertension (systolic blood pressure (BP) >160 mm Hg and/or diastolic BP >100 mm Hg or subjects taking ≥ 2 antihypertensive medications)
* Malignancy
* Current recreational drug or alcohol abuse
* Magnetic resonance imaging (MRI) exclusions: any metal and bio-implants not compatible with 3 Tesla MRI, claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with diabetic ketoacidosis (DKA) will be recruited from Emory University Hospital and Grady Memorial Hospital patients when DKA is treated. Diabetic subjects and age-matched controls will be recruited from physician referrals.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10-25 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Acute change in brain morphology | Baseline, 1 month
  Changes in brain morphology will include quantitative measurements of regional cortical volume as well as of hippocampal and thalamic volumes. Change is the difference from baseline MRI and 1 month MRI.

SECONDARY OUTCOMES:
Long-term change in brain morphology | Baseline, 4 months
  Changes in brain morphology will include quantitative measurements of regional cortical volume as well as of hippocampal and thalamic volumes. Change is the difference from baseline MRI and 4 month MRI.
Change in neurocognitive assessment | Baseline (72 hours after DKA), 3 months
  Assessment will focus in composite domains: verbal memory, visual memory, working memory, prospective memory, executive function processing speed, and reaction time. Change is the difference from baseline assessment and 3 month assessment.
Change in neurocognitive assessment | Baseline (72 hours after DKA), 6 months
  Assessment will focus in composite domains: verbal memory, visual memory, working memory, prospective memory, executive function processing speed, and reaction time. Change is the difference from baseline assessment and 6 month assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Health System, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia